CLINICAL TRIAL: NCT03752619
Title: Peripheral Nerve Stimulation(PNS) for Subacromial Impingement Syndrome(SIS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: University of Texas (Other)
Responsible Party: Principal Investigator, Richard Wilson, MD, Principal Investigator, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB17-00643
Record Dates: First submitted 2018-11-20; First posted 2018-11-26 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Shoulder Pain; Shoulder Impingement Syndrome; Shoulder Tendinitis; Shoulder Bursitis; Pain, Shoulder
Keywords: peripheral nerve stimulation; Sprint; stimulation
MeSH Terms: conditions — Shoulder Pain; Shoulder Impingement Syndrome | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Contraction Producing Peripheral Nerve Stimulation (Experimental): This group will receive: 1) muscle contraction producing peripheral nerve stimulation treatment (which will produce muscle contraction) for three weeks (6 hours daily); and, 2) physical therapy.
  Interventions: Device: Contracting Producing Peripheral Nerve Stimulation; Other: Physical Therapy
- Non Contracting Producing Peripheral Nerve Stimulation (Active Comparator): This group will receive: 1) non contraction producing peripheral nerve stimulation treatment (which will not produce muscle contraction) for three weeks (6 hours daily); and, 2) physical therapy.
  Interventions: Device: Non Contracting Producing Peripheral Nerve Stimulation; Other: Physical Therapy

INTERVENTIONS:
Device: Contracting Producing Peripheral Nerve Stimulation — The stimulation system includes an external stimulator, percutaneous lead and pad. The stimulator snaps onto the pad. The pad has an embedded power source but also serves as the anode. The 1-channel stimulator outputs a biphasic current waveform with current pulse parameter ranges suitable for Peripheral Nerve Stimulation (PNS). The percutaneous lead is inserted using an introducer (like a hypodermic needle) which is withdrawn and the lead is retained in the muscle by a barb at its tip. After a 1-week stabilization period, stimulation is initiated (6 hrs/day). The duty cycle and daily dose remain constant, but stimulus parameters may be adjusted by the research staff as deemed appropriate. The treatment period is 3 weeks after which the lead will be removed.
  Other Names: Intramuscular Peripheral Nerve Stimulation; Intramuscular Electrical Nerve Stimulation; SMARTPATCH System
  Arms: Contraction Producing Peripheral Nerve Stimulation
Device: Non Contracting Producing Peripheral Nerve Stimulation — The stimulation system includes an external stimulator, percutaneous lead and pad. The stimulator snaps onto the pad. The pad has an embedded power source but also serves as the anode. The 1-channel stimulator outputs a biphasic current waveform with current pulse parameter ranges suitable for Peripheral Nerve Stimulation (PNS). The percutaneous lead is inserted using an introducer (like a hypodermic needle) which is withdrawn and the lead is retained in the muscle by a barb at its tip. After a 1-week stabilization period, stimulation is initiated (6 hrs/day). The duty cycle and daily dose remain constant, but stimulus parameters may be adjusted by the research staff as deemed appropriate. The treatment period is 3 weeks after which the lead will be removed.
  Arms: Non Contracting Producing Peripheral Nerve Stimulation
Other: Physical Therapy — All participants receive eight 1.0 hr. sessions of physical therapy (PT) over a 4-wk period from a therapist blinded to Peripheral Nerve Stimulation (PNS) treatment assignment. Each participant also performs home exercises. The primary objective of physical therapy (PT) and the home exercise program is to prevent re-injury by educating and training participants in the biomechanics and proper use of the shoulder and upper limb. During each in-lab session, participants are trained in the implementation of these exercises, which are individually adjusted and progressed with increasing external loads by using weights and elastic rubber bands.

SUMMARY:
Shoulder pain accounts for 16% of all musculoskeletal complaints in the healthy adult population. Subacromial impingement syndrome (SIS) is the most common cause of shoulder pain. Many patients with chronic pain from subacromial impingement syndrome (SIS) will fail treatment efforts and have longstanding pain. This project will evaluate the efficacy of a novel approach to treatment, percutaneous peripheral nerve stimulation, for participants with chronic shoulder pain due to subacromial impingement syndrome (SIS).

DETAILED DESCRIPTION:
The medical and socioeconomic impact of subacute and chronic shoulder pain is high, resulting in 12 million visits to physicians and over $7 billion in direct costs in the United States. The most common cause is subacromial impingement syndrome (SIS), which accounts for 30% of all shoulder pain. Approximately 35% of patients who present with subacromial impingement syndrome (SIS) are refractory to conservative management. For patients who have failed conservative management, there are no established treatments to reduce the pain. The long-term goal is to develop a therapeutic intervention to reduce pain related to subacromial impingement syndrome(SIS). A pilot trial of 3-week percutaneous peripheral nerve stimulation (PNS) for participants with chronic shoulder pain due to subacromial impingement syndrome (SIS) that was refractory to conservative treatment that showed 60% of participants had successful treatment of pain that lasted at least 3 months. Thus, the primary objective of this 2 site randomized control trial (RCT) is to confirm the findings of this preliminary trial and determine the efficacy of peripheral nerve stimulation (PNS) for chronic subacromial impingement syndrome (SIS). The secondary objectives of this multisite randomized control trial (RCT) is to explore mechanisms of peripheral nerve stimulation (PNS) for the treatment of subacromial impingement syndrome (SIS), and to determine which characteristics can predict successful treatment with peripheral nerve stimulation (PNS). In order to accomplish these objectives, this trial is a multi-site, placebo controlled, double-blinded randomized control trial (RCT) to compare the efficacy of peripheral nerve stimulation (PNS) to sham peripheral nerve stimulation (PNS). Measures of pain, pain interference with activities of daily living (ADLs), capacity for activities of daily living (ADLs), Quality of life (QoL), and measures of central sensitization (pain thresholds, secondary hyperalgesia, and temporal summation) will be measured. Participants will be followed for a total of 24 weeks after treatment has concluded.

ELIGIBILITY:
Inclusion Criteria:

1. Shoulder pain of >3 months
2. Age>=21
3. Worst pain in the last week>=4 (0-10 scale)
4. Ability to check skin and perform dressing changes, independently or with assistance
5. Stable dose of pain medication (Not taking more than than 1 opioid or 1 non-opioid analgesic)

Exclusion Criteria:

1. Current shoulder joint or overlying skin infection, or current bacterial infection requiring antibiotics
2. Other chronic pain syndrome (Pain in another area of the body 15 or more days in the last 30 (more than half of the time) or taking daily analgesics for another pain syndrome)
3. Prior shoulder surgery to ipsilateral shoulder joint (glenohumeral, rotator cuff, acromioclavicular (AC) Joint, etc.)
4. Corticosteroid injection in the ipsilateral shoulder or any other pain relieving treatment in last 12 weeks
5. Uncontrolled bleeding disorder
6. Medical instability based on physician opinion after review of medical information
7. Pregnancy
8. Neurological condition affecting ipsilateral upper limb (such as central neurologic injury/illness, radiculopathy, diabetic amyotrophy, Complex Regional Pain Syndrome, etc.)
9. Current Worker's compensation claim for the ipsilateral shoulder
10. Shoulder instability, severe glenohumeral osteoarthritis(OA) based on patient symptoms and physical examination
11. Ipsilateral shoulder injury due to severe trauma (Fall from greater than standing height; Motor vehicle crashes; Struck by vehicle or other fast-moving projectile (e.g., bullet, baseball, etc.); Assault (i.e., injuries intentionally inflicted by another person))
12. Current osseus fracture in ipsilateral arm
13. Ipsilateral upper limb amputation other than a single digit (digits 2-5, partial or full)
14. Surgical indication for shoulder treatment based on physician opinion
15. Compromised immune system (immunodeficiency or immunosuppression)
16. Current use of a Deep Brain Stimulation (DBS) system, implanted active cardiac implant (e.g. pacemaker or defibrillator), any other implantable neuro-stimulator whose stimulus current pathway may overlap with that of the SPRINT System
17. Patients who have a tape or adhesive allergy
18. Contraindication to Magnetic resonance imaging (metal in body, claustrophobia, body habitus, etc) - exclude from Magnetic resonance imaging (MRI) only

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Wilson, MD, Principal Investigator — MetroHealth Medical Center
Locations (2):
- United States (2):
  - MetroHealth Medical Center, Cleveland, Ohio
  - Univerity of Texas Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Urwin M, Symmons D, Allison T, Brammah T, Busby H, Roxby M, Simmons A, Williams G. Estimating the burden of musculoskeletal disorders in the community: the comparative prevalence of symptoms at different anatomical sites, and the relation to social deprivation. Ann Rheum Dis. 1998 Nov;57(11):649-55. doi: 10.1136/ard.57.11.649. PMID 9924205
- [Background] Johnson MP, Crossley KL, O'neil ME, Al-Zakwani IS. Estimates of Direct Health Care Expenditures Among Individuals With Shoulder Dysfunction in the United States J Ortho Sports Phys Ther 2005;35(1,A4).
- [Background] Cadogan A, Laslett M, Hing WA, McNair PJ, Coates MH. A prospective study of shoulder pain in primary care: prevalence of imaged pathology and response to guided diagnostic blocks. BMC Musculoskelet Disord. 2011 May 28;12:119. doi: 10.1186/1471-2474-12-119. PMID 21619663
- [Background] van der Windt DA, Koes BW, de Jong BA, Bouter LM. Shoulder disorders in general practice: incidence, patient characteristics, and management. Ann Rheum Dis. 1995 Dec;54(12):959-64. doi: 10.1136/ard.54.12.959. PMID 8546527
- [Background] Arroll B, Goodyear-Smith F. Corticosteroid injections for painful shoulder: a meta-analysis. Br J Gen Pract. 2005 Mar;55(512):224-8. PMID 15808040
- [Background] Crawshaw DP, Helliwell PS, Hensor EM, Hay EM, Aldous SJ, Conaghan PG. Exercise therapy after corticosteroid injection for moderate to severe shoulder pain: large pragmatic randomised trial. BMJ. 2010 Jun 28;340:c3037. doi: 10.1136/bmj.c3037. PMID 20584793
- [Background] Cummins CA, Sasso LM, Nicholson D. Impingement syndrome: temporal outcomes of nonoperative treatment. J Shoulder Elbow Surg. 2009 Mar-Apr;18(2):172-7. doi: 10.1016/j.jse.2008.09.005. Epub 2008 Dec 18. PMID 19095464
- [Background] Johansson K, Oberg B, Adolfsson L, Foldevi M. A combination of systematic review and clinicians' beliefs in interventions for subacromial pain. Br J Gen Pract. 2002 Feb;52(475):145-52. PMID 11885825
- [Background] Litaker D, Pioro M, El Bilbeisi H, Brems J. Returning to the bedside: using the history and physical examination to identify rotator cuff tears. J Am Geriatr Soc. 2000 Dec;48(12):1633-7. doi: 10.1111/j.1532-5415.2000.tb03875.x. PMID 11129754
- [Background] Morrison DS, Frogameni AD, Woodworth P. Non-operative treatment of subacromial impingement syndrome. J Bone Joint Surg Am. 1997 May;79(5):732-7. doi: 10.2106/00004623-199705000-00013. PMID 9160946
- [Derived] Pierson C, Wilson R, Brewer-Mixon K, Tzen YT, Williamson J, Hansen K, Hisel T, Jain N. Pressure pain sensitivity is independent of structural pathology in patients with subacromial pain syndrome: a cross-sectional analysis. Pain Med. 2025 Apr 1;26(4):173-179. doi: 10.1093/pm/pnae123. PMID 39589920
- [Derived] Cleland T, Jain NB, Chae J, Hansen KM, Hisel TZ, Gunzler DD, Whitehair VC, Kim CH, Wilson RD. The protocol for a multisite, double blind, randomized, placebo-controlled trial of axillary nerve stimulation for chronic shoulder pain. Trials. 2020 Mar 6;21(1):248. doi: 10.1186/s13063-020-4174-x. PMID 32143732
- See also: Functional Electrical Stimulation (FES)Center — http://fescenter.org/index.php
- See also: Metrohealth clinic trials — http://www.metrohealth.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment process at MetroHealth and UTSW included the clinics of the investigators and via referral from the PM&R and orthopedic clinics at each institution. Additionally potential participants were recruited from local area via approved recruitment strategies.
Pre-assignment Details: no pre assignment conditions were used. Subject who met the inclusion and exclusion criteria for the study were enrolled and randomized to a treatment group.
Period: Overall Study
Arm/Group | Contraction Producing Peripheral Nerve Stimulation | Non Contracting Producing Peripheral Nerve Stimulation
Started | 60 | 56
Completed | 57 | 53
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Due to randomization scheme based on baseline characteristics. There are differences in the number of subjects randomized to each group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Contraction Producing Peripheral Nerve Stimulation | Non Contracting Producing Peripheral Nerve Stimulation | Total
Number analyzed (Participants) | 60 | 56 | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 47 | 97
  >=65 years | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years]
  Mean Age | 55.6 (10.39) | 53.2 (13.84) | 54.35 (12.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 27 | 58
  Male | 29 | 29 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 58 | 50 | 108
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 14 | 22
  White | 47 | 38 | 85
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 60 | 56 | 116
Short Form (SF) Question 3 (BPI-SF3) [Mean (Standard Deviation); unit: units on a scale] — Rates pain intensity of the Worst Pain in the last Week on a scale of 0 (no pain) to 10 (worst possible pain).
  units on a scale | 6.90 (1.76) | 7.05 (1.72) | 6.97 (1.75)

OUTCOME MEASURES:

1. Primary Outcome: Change in - Short Form (SF) Question 3 (BPI-SF3)
Description: The Brief Pain Inventory (BPI)has excellent psychometrics. The developers of the Brief Pain Inventory (BPI) recommend Brief Pain Inventory (BPI )3, the "pain worst" rating, as the primary response metric. The question asks participants to rate their worst pain in the prior 24-hours OR prior 7-day on a 0 to 10 Numerical Rating Scale (NRS), where "0" indicates "No pain" and "10" indicates "Pain as bad as you can imagine."
Time Frame: Prior 7-days] ; Baseline (week 1), End of Treatment(week 9), 12 weeks post treatment, 24 weeks post treatment
Population: Numbers of analyzed different between visit due to subject withdrawal, subject compliance.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Contraction Producing Peripheral Nerve Stimulation | Non Contracting Producing Peripheral Nerve Stimulation
Number analyzed (Participants) | 60 | 56
units on a scale
  Baseline(week 1) | 6.90 (1.76) | 7.05 (1.72)
  End of treatment (week 9): number analyzed (Participants) | 60 | 55
  End of treatment (week 9) | 3.58 (2.59) | 3.96 (2.41)
  12 week post treatment: number analyzed (Participants) | 57 | 51
  12 week post treatment | 3.51 (2.90) | 3.53 (2.69)
  24 weeks post treatment: number analyzed (Participants) | 57 | 53
  24 weeks post treatment | 3.04 (2.63) | 3.51 (2.58)

2. Secondary Outcome: Change in Activities of Daily Living(ADL( Capacity - Functional Impairment Test-Hand and Neck/Shoulder/Arm (FIT-HaNSA)
Description: The Functional Impairment Test-Hand and Neck/Shoulder/Arm (FIT-HaNSA) is a laboratory based objective measure of ADL capacity. The Functional Impairment Test-Hand and Neck/Shoulder/Arm (FIT-HaNSA) is a timed test that provides a brief measure of functional ability of the upper limb while performing multi-level tasks that require grip/manipulation of the hand, elbow/shoulder reaching, sustained overhead work, and sustained positioning with an emphasis on assessing the limitations in functional capacity attributable to shoulder and neck disorders.The assessor measures the amount of time that the participant is able to perform each task using a stop watch. The task is completed 3 times- waist level, shoulder level, and eye level. Each task is continued for a maximum of 300 seconds or until a stopping criteria is reached. An overall summary score is calculated by averaging the time for the 3 tasks. Higher numbers indicate higher capacity (range 0-300 seconds).
Time Frame: Baseline (week 1), End of Treatment(week 5), 12 weeks post treatment, 24 weeks post treatment
Population: Numbers of analyzed different between visit due to subject withdrawal, subject compliance.
Measure: Mean (Standard Deviation); unit: Time in seconds
Arm/Group | Contraction Producing Peripheral Nerve Stimulation | Non Contracting Producing Peripheral Nerve Stimulation
Number analyzed (Participants) | 60 | 56
Time in seconds
  Baseline(week 1) | 105.76 (82.76) | 129.95 (75.41)
  End of treatment (week 9): number analyzed (Participants) | 60 | 55
  End of treatment (week 9) | 146.96 (79.27) | 168.32 (83.70)
  12 week post treatment: number analyzed (Participants) | 57 | 52
  12 week post treatment | 140.33 (86.54) | 175.31 (81.13)
  24 weeks post treatment: number analyzed (Participants) | 57 | 53
  24 weeks post treatment | 154.36 (82.88) | 173.61 (76.76)

3. Secondary Outcome: Change in Activities of Daily Living (ADL) Performance -Shoulder Pain and Disability Index (SPADI)
Description: The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The questions ask severity of pain based on an 0-10 numerical Rating Scale where 0 = no pain and 10 = the worst pain imaginable. In addition, it asks how much difficulty the participant has on a numerical rating scale where 0 = no difficulty and 10 = so difficult it requires help. Total disability score: _____/ 80 x 100 = %. Total SPADI score: _____ 130 x 100 = % Higher numbers indicate a higher level of disability (range 0-100%).
Time Frame: Baseline (week 1), End of Treatment(week 5), 12 weeks post treatment, 24 weeks post treatment
Population: Numbers of analyzed different between visit due to subject withdrawal, subject compliance.
Measure: Mean (Standard Deviation); unit: percentage of total disability
Arm/Group | Contraction Producing Peripheral Nerve Stimulation | Non Contracting Producing Peripheral Nerve Stimulation
Number analyzed (Participants) | 60 | 56
percentage of total disability
  Baseline(week 1): number analyzed (Participants) | 60 | 55
  Baseline(week 1) | 48.97 (22.19) | 41.30 (20.57)
  End of treatment (week 9) | 25.78 (22.49) | 21.76 (21.07)
  12 week post treatment: number analyzed (Participants) | 57 | 52
  12 week post treatment | 23.52 (23.64) | 18.88 (21.73)
  24 weeks post treatment: number analyzed (Participants) | 57 | 53
  24 weeks post treatment | 21.90 (22.03) | 20.75 (21.30)

4. Secondary Outcome: Change in Quality of Life - Short Form - 12(QoL - SF 12)
Description: Quality of life - Short form - 12 (QoL - SF 12) is a health related Quality of life (QoL) measure that assesses physical functioning, role limitation because of physical health problems, bodily pain, social functioning, general mental health, role. Scoring: Two summary scores are a mental component score (MCS-12) and a physical component score (PCS-12). The score ranges from 0 - 100 with higher scores indicating better health.
Time Frame: Baseline (week 1), End of Treatment(week 5), 12 weeks post treatment, 24 weeks post treatment
Population: Numbers of analyzed different between visit due to subject withdrawal, subject compliance.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Contraction Producing Peripheral Nerve Stimulation | Non Contracting Producing Peripheral Nerve Stimulation
Number analyzed (Participants) | 60 | 56
units on a scale
  Baseline (week 1) | 38.43 (7.90) | 39.72 (8)
  End of Treatment(week 5): number analyzed (Participants) | 60 | 55
  End of Treatment(week 5) | 44.67 (9.48) | 45.85 (8.56)
  12 weeks post treatment: number analyzed (Participants) | 57 | 52
  12 weeks post treatment | 45.63 (8.56) | 46.39 (9.54)
  24 weeks post treatment: number analyzed (Participants) | 57 | 53
  24 weeks post treatment | 46.97 (9.32) | 46.94 (8.99)

ADVERSE EVENTS:
Time Frame: adverse Event were collected for the time frame subject was enrolled in the study. Eligibility through EOT +6 months, an average of 7 months per participant
Arm/Group | Contraction Producing Peripheral Nerve Stimulation | Non Contracting Producing Peripheral Nerve Stimulation
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/56
Serious Adverse Events (participants affected / at risk) | 2/60 | 5/56
Other Adverse Events (participants affected / at risk) | 40/60 | 35/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Contraction Producing Peripheral Nerve Stimulation (N=60) | Non Contracting Producing Peripheral Nerve Stimulation (N=56)
other Musculoskeletal Injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) — fall, MVA, other pain
other Infection (Infections and infestations) | 0 (0) | 1 (1)
Other Medical condition (Cardiac disorders) | 1 (1) | 1 (1)
Mental Health Concerns (Psychiatric disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Contraction Producing Peripheral Nerve Stimulation (N=60) | Non Contracting Producing Peripheral Nerve Stimulation (N=56)
Skin Irritation (Skin and subcutaneous tissue disorders) | 27 (44) | 21 (32)
Other Musculoskeletal pain/injury (Musculoskeletal and connective tissue disorders) | 13 (15) | 14 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT03752619/Prot_SAP_000.pdf